CLINICAL TRIAL: NCT00916851
Title: Clinical, Environmental, Neurocognitive, Brain Imaging, and Genetic Validity of Autism and Attention-deficit Hyperactivity Disorder
Brief Title: Clinical, Environmental, Neurocognitive, Brain Imaging, and Genetic Validity of Autism and ADHD
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 200903062R
Record Dates: First submitted 2009-06-08; First posted 2009-06-10 (Estimated); Last update posted 2021-09-02 (Actual); Status verified 2021-09

CONDITIONS: Attention Deficit Hyperactivity Disorder; Autism Spectrum Disorder
Keywords: attention-deficit hyperactivity disorder; autism spectrum disorders; normally developing children and adolescents; cognitive functions; emotion/behaviors; brain imaging; genotypes
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Autism Spectrum Disorder; Behavior

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Biospecimen Retention: Samples With DNA — The subjects will receive blood withdrawal. The blood sample will be used for establishing lymphoblastoid cell lines, which will be used for molecular genetic experiments
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Control group: Normally developing children and adolescents
- ADHD group: Children and adolescents with ADHD
- ASD group: Children and adolescents with ASD

SUMMARY:
The behavioral patterns, neurocognitive and social impairments, and high heritability are the common characteristics of autism spectrum disorders (ASD) and attention-deficit hyperactivity disorder (ADHD), the two most common early-onset neuropsychiatric disorders. Little is known about the discriminative validity between these two disorders. As brain imaging studies have been recognized as an important biological tool to validate disease involving the brain, no studies have employed this approach to distinguish the brain functioning between ASD and ADHD. Moreover, there is lack of comprehensive data of environmental, behavioral, neurocognitive, neuroimaging, and genetic data for healthy children. Hence, we propose this program project involving expertise researchers in the fields of child psychiatry and psychology, psychiatric genetics, and brain imaging studies to elucidate the neuropathophysiology and genes & environment interactions of ASD and ADHD as comparing to healthy controls by integrating data from environments, behavioral phenotypes, endophenotypes, and genotypes in one study.

DETAILED DESCRIPTION:
Specific Aims:

1. To compare the individual phenotypes (emotion/behaviors, attention, impulsivity, etc.), endophenotypes (neurocognitive and social cognitive function, brain imaging), and genotypes, and growing environments (prenatal and developmental history, family, school, and social functions) among ASD, ADHD, and normal children to search for etiologies and developmental psychopathologies for ASD and ADHD and to test the discriminative validity of /between ASD and ADHD; and
2. To examine whether the correlations and interactions among/within behavioral phenotypes, endophenotypes, genotypes, and environments vary across the three groups.

This 3-year program project consists of three projects investigating a sample, aged 8-17 years, of 100ASD, 100ADHD, and 100 normally developing children and adolescents.

1. Using diagnostic interviews, observation, self-administered questionnaires, social cognitive tests (emotion recognition test, mentalizing test) and neurocognitive tests (CANTAB, CPT, WCST, WISC-III-R, Émbedded Figure Test, Global-local Perception Test), we will collect data from 300 subjects (100 for each group) regarding individual (phenotype & endophenotype) and growing environments.
2. Using Diffusion Spectrum Imaging, resting-state functional MRI (fMRI), cognitive fMRI (fMRI- semantic association test, fMRI-stroop test), and template, we will collect brain imaging data from 90 subjects regarding individual endophenotype.
3. We will collect the blood samples to establish the cell lines and to conduct SNP genotyping, haplotype, and copy number variation analysis.

With accomplishment of this project, we will not only establish the genotypes for phenotype and endophenotype of general characteristics and assist identifying pathogenesis of ASD and ADHD, but also contribute the etiological studies on several adult psychiatric disorders in future prospective follow-up of this cohort.

ELIGIBILITY:
Inclusion Criteria:

* Control group: Subjects without ADHD or ASD; ADHD group & ASD group: subjects have a clinical diagnosis of ADHD, or ASD defined by the DSM-IV, which was made by a full-time board-certificated child psychiatrist at the first visit and following visits.
* Ages range from 7 to 18 when we conduct the study.
* Subjects have at least one biological parent.
* Both parents are Han Chinese.
* subjects and their biological parents (and siblings if any) consent to participate in this study for complete phenotype assessments and blood withdraw for genetic study

Exclusion Criteria:

* The subjects will be excluded from the study if they currently meet criteria or have a history of the following condition as defined by DSM-IV: Schizophrenia, Schizoaffective Disorder, Organic Psychosis, Mental Retardation, or Pervasive Developmental Disorder. Moreover, the subjects will be excluded from the control group if have a history of the following condition as defined by DSM-IV: ADHD or ASD in addition to the above exclusion criteria.

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: This 3-year program project consists of three projects investigating a sample, aged 8-17 years, of 100 normally developing children and adolescents, 100 ADHD, and 100 ASD.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2010-08-01 (Actual); Primary Completion 2013-07-31 (Actual); Study Completion 2013-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan Shur-Fen Gau, MD, PhD, Principal Investigator — National Taiwan University Hospital & College of Medicine
Locations (1):
- National Taiwan Univeristy Hospital, Taipei, Taiwan

REFERENCES:
- [Derived] Tsai CJ, Lin HY, Tseng IW, Gau SS. White matter microstructural integrity correlates of emotion dysregulation in children with ADHD: A diffusion imaging tractography study. Prog Neuropsychopharmacol Biol Psychiatry. 2021 Aug 30;110:110325. doi: 10.1016/j.pnpbp.2021.110325. Epub 2021 Apr 20. PMID 33857524
- [Derived] Chiang HL, Chen YJ, Shang CY, Tseng WY, Gau SS. Different neural substrates for executive functions in youths with ADHD: a diffusion spectrum imaging tractography study. Psychol Med. 2016 Apr;46(6):1225-38. doi: 10.1017/S0033291715002767. Epub 2016 Jan 8. PMID 26744120
- [Derived] Chiang HL, Chen YJ, Lo YC, Tseng WY, Gau SS. Altered white matter tract property related to impaired focused attention, sustained attention, cognitive impulsivity and vigilance in attention-deficit/ hyperactivity disorder. J Psychiatry Neurosci. 2015 Sep;40(5):325-35. doi: 10.1503/jpn.140106. PMID 25871496